CLINICAL TRIAL: NCT04397016
Title: Cost Talk: a Randomized Stepped Wedge Trial of Interventions Helping Patients Discuss Cancer Care Costs With Clinicians During Shared Decision Making
Brief Title: Cost Talk: Discussing Cancer Care Costs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Robert Wood Johnson Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 202004249
Record Dates: First submitted 2020-05-11; First posted 2020-05-21 (Actual); Last update posted 2022-09-26 (Actual); Status verified 2022-09

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Treatment Costs
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a stepped wedge randomized trial. The intervention condition (the relevant Option Grid decision aid that includes cost information about option) is sequentially assigned to participating surgeons in 4 clusters. By the end of recruitment, all surgeons will have been exposed to the intervention (about 100 surgeon-patient encounters using the Option Grid) and will have provided data for the control (about 100 control cases). Independent eligible patients will be enrolled at each period within a cluster, thus, analyzed as a repeated cross-sectional study. Periods (steps) are set intervals of time. The length of each step is 3 months. Steps 1-3 provide data from both conditions within each cluster (step 0 provides data only from the control while step 4 provides data only from the Option Grid arm) and data is collected from all clusters. Each step will add one clinician to the Option Grid arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Usual Care (No Intervention): * Each participating urologic surgeon will begin in the usual care arm of the study. Subsequently, they will be randomized to the intervention arm at staggered time points to undergo training and begin using the Option Grid decision aid intervention with patients who are diagnosed with slow-growing prostate cancer.
  * Usual Care-Participating clinicians have treatment options discussion with patients with slow-growing prostate cancer. Visits are audio-recorded and/or described by patient self-report measure.
- Arm 2: Option Grid (Experimental): * Each participating urologic surgeon will begin in the usual care arm of the study. Subsequently, they will be randomized to the intervention arm at staggered time points to undergo training and begin using the Option Grid decision aid intervention with patients who are diagnosed with slow-growing prostate cancer.
  * Decision Aid-Participating surgeons use an encounter decision aid to discuss treatment options with patients who have slow-growing prostate cancer. Visits are audio-recorded and/or evaluated by patient self-report measure.
  Interventions: Behavioral: Option Grid Decision Aid

INTERVENTIONS:
Behavioral: Option Grid Decision Aid — -A table with side-by-side comparisons of treatment options organized as responses to patients' frequently asked questions
  Arms: Arm 2: Option Grid

SUMMARY:
The purpose of this study is to investigate whether an encounter decision aid (used during a consultation) containing cost information about options, combined with clinician training about cost discussions and available financial resources, influence surgeon-patient cost conversations, referrals to address costs, patients' financial stress, and high-quality decision-making for patients with slow-growing prostate cancer.

DETAILED DESCRIPTION:
The study will use a stepped wedge design to evaluate the encounter decision aid. Each participating urologic surgeon will begin in the usual care arm of the study. Subsequently, the surgeons will be randomized to the intervention arm at staggered time points to undergo training and begin using the decision aid intervention with patients who are diagnosed with slow-growing prostate cancer. This study will consist of two aims. The first aim is to examine the use of an encounter decision aid with cost information on the presence and impact of out-of-pocket cost conversations. The investigators will train participating clinicians on how to use the decision aid intervention and available financial resources. With patient and clinician consent, the investigators will audio record clinical encounters and measure cost conversations using a previously-developed checklist to code transcripts derived from the audio recordings. Patients can still participate if they do not consent to audio recording as these topics will be assessed in the self-report survey after their clinic or virtual visit. The second aim will examine the impact of an encounter decision aid with cost information on high-quality decision-making. The investigators will collect a post-visit questionnaire from participating patients, including patient-reported measures of decisional conflict, decision regret, and the shared decision-making process. Participants will be sent a follow-up questionnaire 3 months after their initial study enrollment to assess decision regret and financial toxicity.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Visiting a participating urologist/urologic surgeon to discuss treatment options
* Slow growing prostate cancer defined as Gleason score of 6 or 7 (3+4) and/or PSA (prostate-specific antigen) level less than 10ng/ml or at surgeon's discretion
* Must be patients of one of the participating providers

Exclusion Criteria:

-Patients who cannot give informed consent due to cognitive or emotional barriers

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2020-06-12 (Actual); Primary Completion 2022-04-20 (Actual); Study Completion 2022-07-02 (Actual)

PRIMARY OUTCOMES:
Frequency of cost conversations | Immediately after the clinic or virtual visit
Initiator (surgeon, patient, or caregiver) of cost conversations | Immediately after the clinic or virtual visit
Whether or not a referral is made to address costs | Immediately after the clinic or virtual visit

SECONDARY OUTCOMES:
Number of patients who had a decisional conflict | Immediately after the clinic or virtual visit
  The Decisional Conflict Scale assesses whether individuals feel they have enough information to make a choice, have enough support to make a choice, and are clear about their values for risks and benefits of the choice. The 4-item SURE measure of decisional conflict will be used which is scored with a cutoff value indicating whether there is the presence of decisional conflict or not.
Number of patients who engaged in high-quality shared decision-making - CollaboRATE | Immediately after the clinic or virtual visit
  -CollaboRATE is a validated, 3-item measure of the patient's perspective on the level of engagement in their decision. Using the recommended "top score" method of analysis, each encounter is coded as '1', if the response to all three collaboRATE items is 9, or '0' if the response to any of the three collaboRATE items less than 9. Higher scores represent more shared decision making.

OTHER OUTCOMES:
Decision regret | 3 month follow-up
  -The validated Decision Regret Scale consists of five items on a five-point scale from strongly disagree to strongly agree. Higher scores indicate greater decision regret. The investigators will measure regret at the 3-month follow-up and and compare outcomes between groups
Number of patients who had a decisional conflict | 3 month follow-up
  The Decisional Conflict Scale assesses whether individuals feel they have enough information to make a choice, have enough support to make a choice, and are clear about their values for risks and benefits of the choice. The 4-item SURE measure of decisional conflict will be used which is scored with a cutoff value indicating whether there is the presence of decisional conflict or not.
Financial toxicity | 3 month follow-up
  * The investigators will use the validated COST measure of financial toxicity to examine the burden of care costs on patients and their distress about these costs. Higher values indicate more financial toxicity.
  * COST (Comprehensive Score for Financial Toxicity) is a short questionnaire made up of 11 statements. Items are scored on a Likert scale from 0 (not at all) to 4 (very much). Total scores can range from 0 to 44.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Politi, Ph.D., Principal Investigator — Washington University School of Medicine; Glyn Elwyn, M.D., Ph.D., MSc, Principal Investigator — Dartmouth College
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Politi MC, Forcino RC, Parrish K, Durand MA, O'Malley AJ, Moses R, Cooksey K, Elwyn G. The impact of adding cost information to a conversation aid to support shared decision making about low-risk prostate cancer treatment: Results of a stepped-wedge cluster randomised trial. Health Expect. 2023 Oct;26(5):2023-2039. doi: 10.1111/hex.13810. Epub 2023 Jul 2. PMID 37394739
- [Derived] Politi MC, Forcino RC, Parrish K, Durand MA, O'Malley AJ, Elwyn G. Cost talk: protocol for a stepped-wedge cluster randomized trial of an intervention helping patients and urologic surgeons discuss costs of care for slow-growing prostate cancer during shared decision-making. Trials. 2021 Jun 29;22(1):422. doi: 10.1186/s13063-021-05369-4. PMID 34187547
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu